CLINICAL TRIAL: NCT00572221
Title: Improving the Quality of Care in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hebrew SeniorLife (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 06-002; R01NR009071 (NIH); 5R01NR009071-02 (NIH)
Record Dates: First submitted 2007-12-11; First posted 2007-12-12 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Underperforming Nursing Homes
Keywords: CQI; QA; Best Practice; Quality Improvement; Nursing Facilities; Nursing Homes; Care

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- CQI Program Only (Other): The main intervention is a facility-wide Continuing Quality Improvement and Quality Assurance system, with problem recognition and ongoing evaluation. (The SAVE+ intervention, the CQI system with facility responsible for identifying or designing care protocols for the identified problem condition.)
  Interventions: Behavioral: Continuing Quality Improvement and Quality Assurance system
- CQI Program and Best-Practice Care Protocols (Other): A facility-wide Continuing Quality Improvement and Quality Assurance system, with problem recognition and ongoing evaluation. Research clinical staff will also provide best-practice care protocols designed by our research team to address targeted problem conditions. (The SAVE+ intervention, a CQI system plus best-practice protocols designed by study team to address identified problem condition.)
  Interventions: Behavioral: CQI and QA System with Best-Practice Care Protocols

INTERVENTIONS:
Behavioral: Continuing Quality Improvement and Quality Assurance system — The main intervention is a facility-wide Continuing Quality Improvement and Quality Assurance system, with problem recognition and ongoing evaluation.
  Arms: CQI Program Only
Behavioral: CQI and QA System with Best-Practice Care Protocols — A facility-wide Continuing Quality Improvement and Quality Assurance system, with problem recognition and ongoing evaluation. Research clinical staff will also provide best-practice care protocols designed by our research team to address targeted problem conditions.
  Arms: CQI Program and Best-Practice Care Protocols

SUMMARY:
The overall goal of this project is to increase the number of high quality nursing homes in Massachusetts. The study will evaluate an intervention involving two active treatment arms: one implementing a CQI program and a second implementing the CQI program and specific protocol programming. The intervention will be implemented in 24 nursing homes identified as performing, over multiple quality indicator domains, at a poor or average level across multiple outcome domains.

DETAILED DESCRIPTION:
Nursing facilities as well as CMS and state governments are under pressure to find cost-effective methods to improve quality, particularly in poor and average facilities. In our prior work, we found that better performing facilities make more extensive use of CQI mechanisms, have more protocol driven problem advanced resolution mechanisms and systematically address multiple areas Both arms of the study apply the same standardized approach to CQI, while one arm will include specific best-practice care strategies targeted at identified problems. The study will evaluate whether the CQI program improves quality indicator scores in multiple domains, relative to control facilities, and whether improvement is greater in facilities that also utilize the study's best-practice protocols.

The study consent form describes the MDS assessment (used to evaluate the reliability of the facility's assessment), including items to be reviewed and how information will be obtained. The subject is informed that there is no known risk for participating in research, the purpose of which is to determine if the intervention improves nursing home care in Massachusetts

The outcomes will be reviewed by means of a change in twelve quality indicator scores: ADL decline, ADL decline following improvement, Mobility change, walking improvement, cognitive change, communication change, bowel continence change, bladder continence change, depressed mood change, new insertion of an indwelling urinary catheter, infection prevalence, worsening pain.

ELIGIBILITY:
Inclusion Criteria:

* Men and Women
* Residents of long-term care facilities in Massachusetts who have had
* a Minimum Data Set assessment completed by the facility in the last 90 days.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4316 (Actual)
Dates: Start 2006-02; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Change in twelve quality indicator scores | 15 Months

CONTACTS AND LOCATIONS:
Overall Officials: John N Morris, PhD, Principal Investigator — Institute of Aging Research, Hebrew Rehabilitation Center for the Aged
Locations (1):
- Institute for Aging Research, Hebrew Senior Life, Roslindale, Massachusetts, United States